CLINICAL TRIAL: NCT06419140
Title: The Impact of Multimodal Rehabilitation on the Outcomes of Gastric Adenocarcinoma Patients Following Radical D2 Gastrectomy: A Phase II, Multicenter, Open Label, and Randomized Clinical Study
Brief Title: Multimodal Rehabilitation on Gastric Adenocarcinoma Patients Following Radical D2 Gastrectomy
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, Ying Jieer, Chief physician, Zhejiang Cancer Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-2024-349
Record Dates: First submitted 2024-04-16; First posted 2024-05-17 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The rehabilitation group (Experimental): Standard SOX/XELOX adjuvant chemotherapy plus multimodal rehabilitation care
  Interventions: Drug: Standard SOX/XELOX adjuvant chemotherapy plus multimodal rehabilitation
- The control group (No Intervention): Standard SOX/XELOX adjuvant chemotherapy without multimodal rehabilitation care

INTERVENTIONS:
Drug: Standard SOX/XELOX adjuvant chemotherapy plus multimodal rehabilitation — Motivational counseling to perform nutritional, psychological, and exercise inventions
  Arms: The rehabilitation group

SUMMARY:
This study has established a multidisciplinary rehabilitation team to recruit patients who underwent radical D2 gastrectomy in multiple centers and divided them into a rehabilitation group and a control group. Intervention will be carried out every time the patients come to the hospital for adjuvant chemotherapy and review. The control group uses traditional intervention model, and the rehabilitation group uses combined exercise/nutrition/psychology rehabilitation intervention.

This study is expected to promote early recovery after gastric cancer surgery through multidisciplinary rehabilitation intervention, reduce the occurrence of complications, improve patients' tolerance to adjuvant chemotherapy, and improve patients' quality of life, and hope to improve the short-term and long-term outcomes of gastric cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Alzheimer's Disease
* Must be able to swallow tablets
* Age 18 to 75 years old
* Patients with gastric adenocarcinoma (including gastroesophageal junction adenocarcinoma) confirmed by histopathology to be in pathological stage II/III (based on the eighth edition of the AJCC Cancer Staging Manual)
* The patient underwent D2 radical resection within 3-6 weeks before randomization; and met the R0 resection criteria
* The patient can undergo postoperative adjuvant chemotherapy after being selected into the randomization group, and the regimen is SOX/XELOX
* Have not received previous anti-tumor treatment (including systemic chemotherapy and local radiotherapy), except for initial gastrectomy of the primary lesion
* ECOG status score 0 or 1, with physical conditions to participate in sports training、Have sufficient bone marrow reserve function, ANC ≥1.5×109/L, platelet count ≥75×109/L, Hb ≥90 g/L before enrollment, and no bleeding tendency
* Liver function test: alanine aminotransferase (ALT), aspartate aminotransferase (AST), and alkaline phosphatase (ALP) are all ≤ 2.5×ULN; serum bilirubin ≤ 1.5×ULN. For patients known to have Gilbert's disease: Serum bilirubin level ≤ 3ｘULN
* Renal function test: Serum creatinine (Cr) ≤ 1.5 x ULN or creatinine clearance > 50 ml/min (calculated according to Cockroft-Gault)
* No mental illness, speech disorder or consciousness disorder, have certain understanding, communication and reading abilities, and be able to complete the questionnaire independently or with the assistance of the researcher
* During the study, at least one source of social support (family member or friend) can monitor the safety and compliance of the intervention program
* Can understand the situation of this study, and the patient and/or legal representative voluntarily agree to participate in this trial and sign the informed consent form.

Exclusion Criteria:

* Receive neoadjuvant chemotherapy or radiotherapy before surgery;
* Participate in other clinical trials related to health behavior within 3 months before the trial;
* Treated with any other study drugs or participated in another clinical trial with therapeutic intent within 28 days before enrollment;
* Uncontrolled serious medical illness that the investigator believes will affect the subject's acceptance of the rehabilitation program, such as combined serious medical illness, including severe heart disease (such as New York Heart Association (NYHA) Class II or worse congestion heart failure), cerebrovascular disease, uncontrolled diabetes, uncontrolled hypertension, uncontrolled infection, etc.;
* Lack of ability to participate in sports training (such as: disability, paralysis of lower limbs, etc.); not suitable for participating in sports training, such as those suffering from skeletal muscle diseases, fractures within 6 months; suffering from exercise contraindications (angina pectoris, within 6 months) Myocardial infarction, congestive heart failure, chronic obstructive pulmonary disease, planned hip or knee replacement, use of a walker or wheelchair, recent stroke with hemiplegia, etc.);
* Those who are receiving other forms of nutritional intervention; those who refuse to use oral nutritional preparations;
* There is uncontrolled mental illness;
* Known active HIV, HBV and HCV infection;
* Patients with malignant tumors other than gastric cancer (except current gastric cancer) within the past 5 years; are eligible if they meet all the following criteria: treatment of malignant tumors with the purpose of cure, such as fully treated cervical cancer in situ, non-melanoma skin Cancer, localized prostate cancer after radical resection (PSA ≤ 10ng/ml); at the same time, no signs of recurrence or metastasis were found based on imaging follow-up results and any disease-specific tumor markers;
* Those with difficulty swallowing, complete or incomplete gastrointestinal obstruction, active gastrointestinal bleeding, or perforation;
* Pregnant or lactating female patients, or subjects of childbearing age who refuse to take contraceptive measures;
* Patients judged by the researcher to be unfit to participate in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Adjuvant chemotherapy completion rate | At the end of Cycle 8 (each cycle is 21 days)
  Completion rate of 8 cycles of adjuvant chemotherapy

SECONDARY OUTCOMES:
3-year disease-free survival (DFS) | 3 year
  Proportion of subjects who have been free of disease recurrence within 3 years from randomization.
Overall survival | 3 year
  Time from randomization to death
Emotional state | 2 year
  Measured by GAD-7 questionnaire
Weight | through study completion, an average of 2 year
  Weight
Adverse event | At the end of Cycle 8 (each cycle is 21 days)
  Adverse event were evaluated through CTCAE

CONTACTS AND LOCATIONS:
Overall Officials: Jieer Jieer, Dr, Principal Investigator — Zhejiang Cancer Hospital
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No